CLINICAL TRIAL: NCT05431218
Title: Association of Cathelicidin and Vitamin D Levels With the Category and Course of COPD
Acronym: COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karaganda Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VitD COPD
Record Dates: First submitted 2022-05-25; First posted 2022-06-24 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Chronic Obstructive Pulmonary Disease; Chronic Obstructive Pulmonary Disease Moderate; Chronic Obstructive Pulmonary Disease Severe
Keywords: COPD; vitamin D; cathelicidin; antimicrobial peptide
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: The study suggests dividing patients, depending on the initial vitamin D level, into 4 groups: normal level, deficiency, deficiency and severe deficiency. Also, the division into groups according to the severity of chronic obstructive pulmonary disease: mild, moderate, severe and extremely severe
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- normal vitamin D levels (No Intervention): Patients with normal vitamin D levels (30-100ng/ml) No interference is implied. Observation only
- Mild vitamin D deficiency (Active Comparator): Patients with mild vitamin D deficiency (20-29 ng/ml)They will receive 4000 IU of cholecalciferol per day for 3 months
  Interventions: Drug: Cholecalciferol Liquid
- Moderate vitamin D deficiency (Active Comparator): Patients with moderate vitamin D deficiency (10-19 ng/ml) will receive cholecalciferol at a dose of 5000-6000 IU daily for 3 months
  Interventions: Drug: Cholecalciferol Liquid
- Severe vitamin D deficiency (Active Comparator): Patients with moderate vitamin D deficiency (10-19 ng/ml) will receive cholecalciferol at a dose of 7000-8000 IU daily for 3 months
  Interventions: Drug: Cholecalciferol Liquid

INTERVENTIONS:
Drug: Cholecalciferol Liquid — daily single dose of the drug in the first half of the day in an individually selected dose for 3 months
  Other Names: D vitamin
  Arms: Mild vitamin D deficiency; Moderate vitamin D deficiency; Severe vitamin D deficiency

SUMMARY:
Recruitment of patients with COPD. Assessment of clinical status, determination of vitamin D and cathelicidin levels. In the group with vitamin D deficiency, patients receive cholecalciferol (vitamin D) daily for 3 months. After 3 months, the clinical status was assessed again, the level of vitamin D and cathelicidin was determined. When vitamin D levels normalize, cholecalciferol replacement therapy is discontinued for 3 months. After that, a control inspection and laboratory tests are performed.

DETAILED DESCRIPTION:
Interventional prospective research design.

The study will be conducted on patients with moderate and severe COPD. The material for the study will be the blood and sputum of patients with COPD.

Research methods: biochemical, enzyme immunoassay, bacteriological, radiological, spirography, clinical, statistical analysis.

The recruitment of patients is carried out in the pulmonology department of the hospital according to the inclusion and exclusion criteria. Patient participation is voluntary. First, the patient is told about the study. If he agrees, he signs an informed consent to conduct research.

Clinical examination of the patient, anthropometry, standard COPD assessment tests will be conducted in the hospital.

Laboratory tests will be conducted in medical institutions in Karaganda and will include a detailed general blood test, determination of fibrinogen and CRP (C-reactive protein) levels, general sputum analysis and bacteriological sputum examination.

Instrumental studies are carried out in medical institutions of the city: spirometry (determination of FEV1 (forced exhalation volume), Gensler index and Tiffno), lung radiography.

The study of vitamin D and cathelicidin is carried out by the ELISA method in the laboratory of the Medical University. Assessment of vitamin D status will be carried out by determining the level of total 25(OH)D (circulating serum, total D2 and D3) with verification of the method relative to international standards (National Institute of Standards and Technology - National Institute of Standards and Technology (NIST), Vitamin D External Quality Assessment Scheme (DEQAS)). The interpretation of vitamin D levels will be carried out according to international standards:

less than 10 ng/ml severe deficiency; 10-20 ng/ml moderate deficiency; 20-30 ng/ml mild deficiency; 30-100 ng/ml Norm; more than 100 ng/ml toxic level.

Quantitative determination of the level of antimicrobial peptide cathelicidin (LL-37) in blood serum will be carried out using enzyme immunoassay (NK321, HumanLL-37 ELISA Kit, Hycult biotech, the Netherlands) in accordance with the manufacturer's instructions. . Normal levels of LL-37: 50-80 ng/ml.

Among the patients with COPD selected at the outpatient stage, persons with vitamin 25(OH) deficiency were identifiedD in the blood (insufficiency/deficiency). In this group, patients received a therapeutic dose of an aqueous solution of cholecalciferol for three months. The therapeutic dose of an aqueous solution of cholecalciferol will be calculated individually according to clinical recommendations for the treatment of vitamin D deficiency and insufficiency.

Patients will continue treatment of the underlying COPD disease according to the clinical protocol. Vitamin therapy is an addition to the main treatment, it should strengthen the immunity and protective abilities of the body. After three months of replacement therapy with cholecalciferol and the next 3 months without it, clinical, laboratory and instrumental research methods will be repeated to assess the effectiveness.

Statistical processing of the research results is supposed to be carried out using statistical packages Excel 2010 (Microsoft, USA), Statistica 10.0 (StatSoft, Inc., USA). Methods of parametric and nonparametric statistics will be used: Student's criterion (t), Mann-Whitney (U), Wilcoxon; correlation analysis with calculation of Spearman's correlation coefficient (R). To compare the case-control groups with a quantitative assessment of the relationship between the factor and the outcome, the odds ratio (OR) with 95% CI will be calculated.

ELIGIBILITY:
Inclusion Criteria:

- Clinically confirmed chronic obstructive pulmonary disease

Exclusion Criteria:

* age under 18
* pregnancy
* mental disorders
* cancer
* terminal renal and hepatic insufficiency

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Dynamics of vitamin D levels at baseline and 3 months | At baseline and 3 months
  Assessment of the levels of vitamin D (ng / ml) in blood plasma and evaluate the dynamics of the measurement of the indicator in the same patient in different periods of time, and compare the indicators in groups of patients
Dynamics of vitamin D levels at baseline and 6 months | At baseline and 6 months
  Assessment of the levels of vitamin D (ng / ml) in blood plasma and evaluate the dynamics of the measurement of the indicator in the same patient in different periods of time, and compare the indicators in groups of patients
Dynamics of vitamin D levels at 3 months and 6 months | At 3 months and 6 months
  Assessment of the levels of vitamin D (ng / ml) in blood plasma and evaluate the dynamics of the measurement of the indicator in the same patient in different periods of time, and compare the indicators in groups of patients
Dynamics of cathelicidin levels at baseline and 3 months | At baseline and 3 months
  Assessment of cathelicidin levels (ng / ml) in blood plasma and and evaluate the dynamics of the measurement of the indicator in the same patient in different periods of time, and compare the indicators in groups of patients
Dynamics of cathelicidin levels at baseline and 6 months | At baseline and 6 months
  Assessment of cathelicidin levels (ng / ml) in blood plasma and and evaluate the dynamics of the measurement of the indicator in the same patient in different periods of time, and compare the indicators in groups of patients
Dynamics of cathelicidin levels at 3 months and 6 months | At 3 months and 6 months
  Assessment of cathelicidin levels (ng / ml) in blood plasma and evaluate the dynamics of the measurement of the indicator in the same patient in different periods of time, and compare the indicators in groups of patients

CONTACTS AND LOCATIONS:
Locations (1):
- Karaganda Medical University, Karaganda, Kazakhstan

REFERENCES:
- See also: Uysal P, Simsek G, Durmus S, Sozer V. Evaluation of plasma antimicrobial peptide LL-37 and nuclear factor-kappaB levels in stable chronic obstructive pulmonary disease 25 January 2019 Volume 2019:14 Pages 321-330 — https://pubmed.ncbi.nlm.nih.gov/30774329/
- See also: World Health Organization official website — http://www.who.int
- See also: International conference "Respiratory Junction Almaty: Where East meets West". 02.04.2019 — http://www.kaznu.kz/ru/20215/news/one/16350/
- See also: Yang YM, Guo YF, Zhang HS, Sun TY. Antimicrobial peptide LL-37 circulating levels in chronic obstructive pulmonary disease patients with high risk of frequent exacerbations. J Thorac Dis. 2015;7(4):740-745 — http://www.ncbi.nlm.nih.gov/pubmed/25973241
- See also: V. Casanova, F.H. Sousa, C. Stevens, P. Barlow Antiviral therapeutic approaches for human rhinovirus infections Future Virol., 13 (2018), pp. 505-518 CrossRefView Record in ScopusGoogle Scholar — http://www.ncbi.nlm.nih.gov/pubmed/30245735
- See also: Roby KD, Nardo AD. Innate immunity and the role of the antimicrobial peptide cathelicidin in inflammatory skin disease. Drug Discov Today Dis Mech. 2013;10(3-4):e79-e82. doi:10.1016/j.ddmec.2013.01.001 — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3904447/
- See also: Burkes RM, Astemborski J, Lambert AA, et al. Plasma cathelicidin and longitudinal lung function in current and former smokers. PLoS One. 2019;14(2):e0212628. Published 2019 Feb 27. doi:10.1371/journal.pone.0212628 — http://www.ncbi.nlm.nih.gov/pubmed/30811465
- See also: Vitamin D Supplement Doses and Serum 25-Hydroxyvitamin D in the Range Associated with Cancer Prevention C.F. GARLAND, C.B. FRENCH, L.L. BAGGERLY and R.P. HEANEY Anticancer Research February 2011 vol.31 no.2 6007-611 — https://pubmed.ncbi.nlm.nih.gov/21378345/